CLINICAL TRIAL: NCT05999539
Title: Comparison of Demography, Functional Capacity, Prosthesis Type and Health-related Quality of Life Between Faller and Non-faller Transtibial Amputees
Brief Title: Comparison of Characteristics Between Faller and Non-faller Transtibial Amputees
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Yasin YURT, Assoc. Prof. Dr., Eastern Mediterranean University
Other Study IDs: ETK00-2023-0130
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Amputation; Fall; Ambulation Difficulty; Quality of Life; Prosthesis User
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Faller transtibial prosthetic users: Transtibial prosthetic users who fell at least once in the last year.
  Interventions: Device: Transtibial prosthesis
- Non-faller transtibial prosthetic users: Transtibial prosthetic users who have no fall history.
  Interventions: Device: Transtibial prosthesis

INTERVENTIONS:
Device: Transtibial prosthesis — A transtibial prosthesis to be used for at least one year.

SUMMARY:
Researchers aim to compare demographic characteristics, prosthesis type, functional capacity, and quality of life between faller and non-faller transtibial amputees.

DETAILED DESCRIPTION:
Unilateral transtibial level prosthetic users will be included in this study. After getting the fall history of subjects, those who feel at least one time or more in the last year will be accepted as the faller group. Demographic characteristics, functional capacity, health-related quality of life, and prosthetic types used by amputees will be assessed. The main differences between the faller and non-faller transtibial amputees will be analyzed with the data.

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to walk at least 30-meter independently
* Using the transtibial prosthesis for at least one year.

Exclusion Criteria:

* Multiple limb amputees or prosthetic users
* Having prosthetic discomfort or stump ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be the transtibial prosthetic users recorded in outpatient clinics working on amputee rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Two-minute walk test | 1 week
  The test to be carried out to find out functional capacity, in a 30-meter-long area will be marked at 3-meter intervals, and the turning points will be determined with an object such as a traffic cone. We will ask the individual to walk the maximum distance in 2 minutes and we will tell them that they can slow down and stop when they get tired. When 2 minutes are completed with a stopwatch, we will ask the individual to stop and record the walking distance in meters.

SECONDARY OUTCOMES:
Functional Reach Test | 1 week
  This test will be used to assess balance. The subjects will be asked to stand sideways next to the wall and wait with the shoulder in 90 degrees flexion, elbow in extension and fist closed without touching the wall with the arm close to the wall. The 3rd metacarpal head will be marked and the patient will be asked to reach as far as they can without taking a step, then the new location of the 3rd metacarpal head will be marked. Scoring will be determined by measuring the difference between the start and end position in centimeters. 3 attempts will be made and the best result will be taken.
Timed Up and Go Test | 1 week
  This test will be used to assess fall risk. A distance of 3 meters will be determined in front of the chair, the individual is asked to get up from the chair and walk the determined distance, and the time elapsed will be recorded with a stopwatch with seconds.
Trinity Amputation and Prosthesis Experiences Scales | 1 week
  This test is used to assess different aspects of amputees' experience of prosthesis use and quality of life. It gives a total score that means better when higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data of participants will not be shared individually because of health policy. Results will be shared as an overall data.